CLINICAL TRIAL: NCT01711515
Title: A Phase I Trial of Sequential Ipilimumab After Chemoradiation for the Primary Treatment of Patients With Locally Advanced Cervical Cancer Stages IB2/IIA With Positive Para-Aortic Lymph Nodes Only and Stage IIB/IIIB/IVA With Positive Lymph Nodes
Brief Title: Chemoradiation Therapy and Ipilimumab in Treating Patients With Stages IB2-IIB or IIIB-IVA Cervical Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01733; NCI-2012-01733 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-PIS1102; GOG-9929; GOG-9929 (Other: NRG Oncology); GOG-9929 (Other: CTEP); U10CA180830 (NIH); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma, Not Otherwise Specified; Stage IB2 Cervical Cancer AJCC v6 and v7; Stage II Cervical Cancer AJCC v7; Stage IIA Cervical Cancer AJCC v7; Stage IIB Cervical Cancer AJCC v6 and v7; Stage IIIB Cervical Cancer AJCC v6 and v7; Stage IVA Cervical Cancer AJCC v6 and v7
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Radiation; Brachytherapy; Ipilimumab; CTLA-4 Antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (cisplatin, radiation therapy, and ipilimumab) (Experimental): Patients receive cisplatin IV over 1 hour on days 1, 8, 15, 22, 29, and 36, undergo extended beam radiation therapy 5 days a week for 6 weeks, and then undergo intracavitary brachytherapy for approximately 2 weeks. Within 2 weeks, patients receive ipilimumab IV over 90 minutes once every 3 weeks for 12 weeks.
  Interventions: Drug: Cisplatin; Radiation: External Beam Radiation Therapy; Radiation: Internal Radiation Therapy; Biological: Ipilimumab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone''s Chloride; Peyrone''s Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Radiation: External Beam Radiation Therapy — Undergo external beam radiation therapy
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam
Radiation: Internal Radiation Therapy — Undergo intracavitary brachytherapy
  Other Names: Brachytherapy; Brachytherapy, NOS; Internal Radiation; Internal Radiation Brachytherapy; Radiation Brachytherapy; Radiation, Internal
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of ipilimumab when given after chemoradiation therapy in treating patients with stages IB2-IIB or IIIB-IVA cervical cancer. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Monoclonal antibodies, such as ipilimumab, may find tumor cells and help carry tumor-killing substances to them. Giving ipilimumab together with chemoradiation therapy may be a better way treat cervical cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and dose-limiting toxicities (DLT) of adjuvant ipilimumab following concurrent weekly cisplatin and extended field radiation in women with newly diagnosed locally advanced cervical cancer stage IB2/ IIA with-positive para-aortic lymph nodes only and stage IIB/IIIB/IVA with positive lymph nodes.

II. To determine the feasibility of the treatment regimen over the four cycles of adjuvant ipilimumab once the MTD is estimated.

III. To assess the toxicities of the treatment regimen per the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

SECONDARY OBJECTIVES:

I. To examine progression free survival for 1 year after study completion. II. To determine site of recurrence, loco-regional versus distant, for one year after completion of therapy.

III. To estimate the frequency of chronic toxicities experienced within one year after completion of therapy.

TERTIARY OBJECTIVES:

I. To enumerate the human papillomavirus (HPV)-subtype-specific T-cells and characterize the kinetics of HPV-subtype-specific T-cell expansion associated with chemoradiation and ipilimumab treatment.

II. To characterize the association between differential expression of immune markers on leukocytes from human leukocyte antigen (HLA)-A*0201 patients and response to chemoradiation and ipilimumab treatment.

III. To assess qualitative changes in maximum standardized uptake value (SUVmax) from positron emission tomography (PET)/computed tomography (CT) after treatment with chemoradiation and ipilimumab.

IV. To bank residual plasma (obtained from leukocyte processing) for future research.

OUTLINE: This is a dose-escalation study of ipilimumab.

Patients receive cisplatin intravenously (IV) over 1 hour on days 1, 8, 15, 22, 29, and 36, undergo external beam radiation therapy 5 days a week for 6 weeks, and then undergo intracavitary brachytherapy for approximately 2 weeks. Within 2 weeks, patients receive ipilimumab IV over 90 minutes once every 3 weeks for 12 weeks.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed advanced cervical cancer (squamous cell carcinoma, adenocarcinoma, and adenosquamous cell carcinoma): International Federation of Gynecology and Obstetrics (FIGO) clinical stages IB2/IIA with positive para-aortic lymph nodes or FIGO clinical stages IIB/IIIB/IVA with positive pelvic and/or para-aortic lymph nodes; nodal status will be confirmed by PET/CT scan, fine needle biopsy, extra peritoneal biopsy, laparoscopic biopsy or lymphadenectomy
* Patients must have a Gynecologic Oncology Group (GOG) performance status of 0-1
* Absolute neutrophil count (ANC) >= 1,500/mcl
* Platelets >= 100,000/mcl
* Creatinine =< institutional upper limit normal (ULN); note: if creatinine > ULN, creatinine clearance must be > 50 mL/min
* Bilirubin =< 1.5 x ULN
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN
* Alkaline phosphatase =< 2.5 x ULN
* Neuropathy (sensory and motor) =< grade 1
* Patients with ureteral obstruction (i.e., hydronephrosis identified on CT imaging) must undergo stent or nephrostomy tube placement prior to study entry
* Patients must meet the pre-entry requirements specified
* Patients must have signed an approved informed consent and authorization permitting the release of personal health information
* Patients of child-bearing potential must have a negative serum pregnancy test prior to study entry (within 72 hours prior to initiation of study treatment) and be practicing an effective form of contraception; women should not breast-feed while on this study
* Patients must not be receiving any other investigational agent
* Patients should have an audiogram at baseline, and patients with pre-existing hearing loss or hearing loss during treatment should be assessed frequently during cisplatin therapy

Exclusion Criteria:

* Patients who have received previous pelvic or abdominal radiation, cytotoxic chemotherapy, or previous therapy of any kind for this malignancy or any pelvic or abdominal radiation for any prior malignancy
* Patients with active infection
* Patients who have circumstances that will not permit completion of this study or the required follow-up
* Patients with renal abnormalities, such as pelvic kidney, horseshoe kidney, or renal transplantation, that would require modification of radiation fields
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last five years; patients are also excluded if their previous cancer treatment prevents full delivery of this protocol therapy
* Patients who have undergone major surgery, excluding diagnostic biopsy, within 30 days (to allow for full recovery) prior to registration
* Patients who have a significant history of cardiac disease, i.e., uncontrolled hypertension, unstable angina, congestive heart failure, or uncontrolled arrhythmias within 6 months of registration
* Patients with a history of prior treatment with ipilimumab, anti-programmed cell death (PD) 1 antibody, cluster of differentiation (CD)137 agonist or other immune activating therapy such as anti-CD 40 antibody
* Patients who are receiving any other investigational agents
* Autoimmune disease: patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's disease, are excluded from this study, as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis]); central nervous system (CNS) or motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre syndrome and myasthenia gravis, multiple sclerosis)
* Patients with known immune impairment who may be unable to respond to anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA 4) antibody
* History of allergic reactions attributed to compounds of similar chemical or biologic composition ipilimumab or other agents used in study
* Patients with chronic human immunodeficiency virus (HIV), hepatitis B or hepatitis C infections should be excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
DLTs occurring during adjuvant ipilimumab in the dose escalation phase | During first 2 courses of treatment
DLTs occurring in the feasibility phase | Over 4 courses of treatment
Toxicities as assessed by CTCAE version 4 | Up to 2 years post-treatment

SECONDARY OUTCOMES:
Response rate in patients enrolled with measurable disease assessed using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Up to 2 years post-treatment
  Relationships of translational research endpoints to response will be explored if practical.
Progression-free survival (PFS) | From time of study entry to time of progression or death, whichever occurs first, assessed up to 1 year post-treatment
  Will be summarized using Kaplan-Meier plots. Relationships of translational research endpoints to PFS will be explored if practical.
Overall survival | From time of study entry to time of death or the date the patient was last confirmed to be alive, assessed up to 1 year post-treatment
  Will be summarized using Kaplan-Meier plots.
Location of recurrence (loco-regional versus distant) | Up to 1 year post-treatment
Chronic toxicities experienced within one year of completion of therapy | Up to 1 year post-treatment

OTHER OUTCOMES:
Enumeration of HPV-specific T-cells | Up to 2 years
  Summary statistics (and graphs) of translational research endpoints will be done by dose level. Relationships of these endpoints to response and PFS will be explored if practical.
Kinetics of HPV-specific T-cell expansion | Up to 2 years
  Summary statistics (and graphs) of translational research endpoints will be done by dose level. Relationships of these endpoints to response and PFS will be explored if practical.
Characterization of differential activated T-cell responses based on HLA-subtype A*0201 | Up to 2 years
  Summary statistics (and graphs) of translational research endpoints will be done by dose level. Relationships of these endpoints to response and PFS will be explored if practical.
Measurable parameters from the fludeoxyglucose F 18 (FDG)-PET/CT, including SUVmax of the primary tumor, metabolic tumor volume (MTV) if available, the presence of abnormal FDG uptake within lymph nodes | Up to 2 years
  Summary statistics (and graphs) of translational research endpoints will be done by dose level. Relationships of these endpoints to response and PFS will be explored if practical. Within-patient changes in the FDG-PET/CT SUVmax and MTV (if available) will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti S Mayadev, Principal Investigator — NRG Oncology
Locations (16):
- United States (16):
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Augusta University Medical Center, Augusta, Georgia
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Derived] Da Silva DM, Enserro DM, Mayadev JS, Skeate JG, Matsuo K, Pham HQ, Lankes HA, Moxley KM, Ghamande SA, Lin YG, Schilder RJ, Birrer MJ, Kast WM. Immune Activation in Patients with Locally Advanced Cervical Cancer Treated with Ipilimumab Following Definitive Chemoradiation (GOG-9929). Clin Cancer Res. 2020 Nov 1;26(21):5621-5630. doi: 10.1158/1078-0432.CCR-20-0776. Epub 2020 Aug 18. PMID 32816895